CLINICAL TRIAL: NCT03676634
Title: Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers With Existing Botulinum Immunity
Brief Title: Tolerability and Immunogenicity of rBV A/B for the Production of BabyBIG®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Department of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: rBV A/B-CL-002
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2020-01

CONDITIONS: Botulism
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental): rBV A/B
  Interventions: Biological: rBV A/B

INTERVENTIONS:
Biological: rBV A/B — Recombinant Botulinum Vaccine A/B, rBV A/B

SUMMARY:
This Phase 2, open-label, uncontrolled study designed to evaluate safety, tolerability, and immunogenicity of a single dose of rBV A/B in healthy participants previously immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection will be conducted to collect source plasma for potential use in the production of BabyBIG and to evaluate safety and immunogenicity of the vaccine in these participants over a 12-week period, with a follow-up safety assessment at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have received pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection under BB IND 0161 (or BB-IND-0161 and IND 015155)
2. Be 18 to 69 years old at the time of consent
3. Be healthy and have an acceptable medical history that will not interfere with the objectives of the study
4. Meet the participant suitability requirements and recommendations for source plasma donors outlined in Appendix A.
5. If female, and of childbearing potential, have a negative pregnancy test at screening and within 24 hours prior to vaccination and must not plan to become pregnant until after the last plasma donation or until the Week 12 visit ([whichever occurs last].
6. Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by the Committee for the Protection of Human Subjects, and have agreed to abide by the study restrictions and to return for the required assessments
7. Agree to complete the participant home diary on a daily basis for 7 days post vaccination, as well as to report any adverse events and concomitant medications during the study period
8. Have provided written authorization for use and disclosure of protected health information
9. Agree not to donate blood or blood products (outside of study procedures) until after the last plasma donation or until the Week 12 visit (whichever occurs last)
10. Have personal health insurance

Exclusion Criteria:

1. Be pregnant or nursing
2. Have a history of laboratory evidence of syphilis, acquired immunodeficiency syndrome, Creutzfeldt-Jakob disease, or infection with human immunodeficiency viruses (HIV) 1 or 2, human T-cell lymphotropic virus 1, hepatitis B virus (HBV), or hepatitis C virus (HCV)
3. Have had a prior severe (Grade 3 or higher) local or severe (Grade 3 or higher) systemic reaction to last immunization with pentavalent botulinum toxoid or a prior severe immediate hypersensitivity reaction or severe systemic reaction to last vaccination on Day 0 with rBV A/B
4. Have known allergy to aluminum, yeast, or other components of the vaccine
5. Have donated one or more units of blood or undergone plasmapheresis within 49 days of the Vaccination Visit (Day 0)
6. Have received blood product or immunoglobulin within 6 months prior to study entry or plans to receive such products during the study period (exclusive of returned red blood cells as part of the plasmapheresis procedure). For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
7. Have received licensed nonliving vaccine within 14 days prior to study entry, or licensed live vaccine within 60 days prior to study entry
8. Have received investigational products (drugs, biologics, vaccines, or implantable devices) 60 days prior to study entry or plans to receive experimental products at any time during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
9. Have received prescription immunosuppressive or immunomodulatory agents, including parenteral, inhaled, or oral corticosteroids within 3 months of study entry or plans on receiving such therapy at any time during the study period [For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)], with the exceptions mentioned below

   * Participants who have used prescription topical steroids may be enrolled 2 weeks after the therapy is completed
   * Intra-articular, bursal, or tendon injectable steroids are permitted
   * Any over-the-counter topical steroid use is permitted
   * Ophthalmic and intranasal steroids are permitted
10. Have received cytotoxic therapy at any time in the previous 5 years before study entry
11. Have an active systemic or recurrent disease that would place the participant at unacceptable risk of injury, require hospitalization, or require surgical intervention (This includes active mental illness or history of mental illness not responsive to treatment.)
12. Have a history of alcohol or drug abuse or dependence within 12 months of study entry
13. Have past, present, or suspected illicit injection drug use
14. Have inflammatory, vasculitic, or rheumatic disease, including systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma (Stable osteoarthritis treated with physical therapy and nonsteroidal anti inflammatory drugs is not an exclusion criterion.)
15. Have any acute or chronic neuromuscular or neurologic disorder
16. Have clinically confirmed hepatic or renal insufficiency
17. Have uncontrolled hypertension, as defined a systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 90 mmHg
18. Have moderate to severe asthma, chronic obstructive pulmonary disease, or other significant pulmonary disease
19. Have a seizure disorder
20. Have moderate or severe illness or oral temperature of 100.4°F or greater within 3 days of Vaccination Visit (Day 0)
21. Be unsuitable for participation in this study for any reason, as assessed by the investigator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Arnon, M.D., M.P.H., Principal Investigator — California Department of Public Health
Locations (2):
- United States (2):
  - California Department of Public Health, Richmond, California
  - Battelle Biomedical Research Center, West Jefferson, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants were enrolled during the recruiting period from 07 March 2019 to 29 August 2019.
Pre-assignment Details: All enrolled participants participated in the study.
Groups:
- 0.5 mL rBV A/B: A single 0.5-mL intramuscular injection of 40 μg of rBV A/B was administered to each participant on Day 0 to stimulate the production of antibodies against botulinum toxin type A and type B.
Period: Overall Study
Arm/Group | 0.5 mL rBV A/B
Started | 32
Screening | 32
Participants Received rBV A/B Injection | 32
Participants Included in the Plasma-donating Population | 32
Participants Completed Follow up | 32
Completed | 29
Not Completed | 3
Not completed — Red blood cell loss | 1
Not completed — Out-of-limit pulse | 2

BASELINE CHARACTERISTICS:
Arm/Group | 0.5 mL rBV A/B
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.80)
Age, Continuous [Median (Full Range); unit: years] | 44.5 [33 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
Previous BabyBIG Plasma Donor [Number; unit: participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Greater Than 3- or 4-Fold Increases in Neutralizing Antibody Concentration (NAC)
Description: Neutralizing Antibody Concentration in Plasma
Time Frame: Week 0 to Week 4
Population: Immunogenicity Population: All participants who received rBV A/B, had a baseline NAC, and had at least one post-vaccination immunogenicity assessment up to and including four weeks after administration of rBV A/B
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.5 mL rBV A/B
Number analyzed (Participants) | 32
proportion of participants
  Proportion of participants with a ≥4x increase in type A NAC | .844 [.672 to .947]
  Proportion of participants with a ≥3x increase in type A NAC | .938 [.792 to .992]
  Proportion of participants with a ≥4x increase in type B NAC | .875 [.710 to .965]
  Proportion of participants with a ≥3x increase in type B NAC | .906 [.750 to .980]
Statistical Analysis 1: Comparison: 0.5 mL rBV A/B; Consider increase from baseline to post-dose values. Parameter is proportion achieving desired increase (≥ 3x or 4x increase in Type A and Type B NAC); Test type: Other; single proportion = .844, 95% CI 2-sided [.672 to .947] — Values listed in table are for Type A. Estimated Value for the Estimation Parameter for type B = 0.875. Lower limit = 0.710, upper limit = 0.965; Proportion of participants achieving ≥ 3x or 4x increase in NAC values was calculated for both Type A and Type B. Primary endpoint was achieved if both Type A and Type B had proportion ≥50%

2. Secondary Outcome: Proportion of Subjects Achieving Greater Than 2-Fold Increase in Neutralizing Antibody Concentration (NAC)
Description: Neutralizing Antibody Concentration in Plasma
Time Frame: Week 0 to 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.5 mL rBV A/B
Number analyzed (Participants) | 32
proportion of participants
  two times or greater increase in type A NAC compared with Week 0 | .906 [.750 to .980]
  two times or greater increase in type B NAC compared with Week 0 | .844 [.672 to .947]

3. Other Pre Specified Outcome: Volume of Plasma Collected With an Acceptable Anti-type A or Anti-type B Titer
Description: Neutralizing Antibody Concentration in Plasma
Time Frame: Week 0 to 4
Population: Plasma-Donating Population: all participants who received rBV A/B and donated at least one plasma unit.
Measure: Number; unit: mL
Arm/Group | 0.5 mL rBV A/B
Number analyzed (Participants) | 32
mL
  Total volume of plasma from all donating participants | 470,102
  Total volume of plasma from donating participants with any positive titer | 470,102
  Total volume of plasma from donating participants with positive anti-A titer | 470,102
  Total volume of plasma from donating participants with positive anti-B titer | 469,411

ADVERSE EVENTS:
Time Frame: Non-serious AEs (injection site reactions/systemic reactions) were only collected from day 0 - day 7 during the participant diary collection period. For the rest of the study (from day 7 through 12 weeks of site visits and through the week 26 follow up phone call), AEs were only collected if they were SAEs.
Description: Mortality, Adverse Events, and Serious Adverse Event definitions are as described on clinicaltrials.gov. Any anticipated or unanticipated events (not included in the serious adverse event table) grouped by organ system, with the number and frequency of such events.
Arm/Group | 0.5 mL rBV A/B
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 5/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mL rBV A/B (N=32)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mL rBV A/B (N=32)
injection site erythema (General disorders) | 4 (4) — general disorders and administration site conditions
injection site induration (General disorders) | 3 (3) — general disorders and administration site disorders
injection site pain (General disorders) | 1 (1) — general disorders and administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT03676634/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03676634/SAP_001.pdf